CLINICAL TRIAL: NCT04046848
Title: Phase 1/2 Study to Assess the Safety and Pharmacokinetics of Subcutaneous Injection of OCTA101 in Previously Treated Adult Patients With Severe Hemophilia A
Brief Title: Safety and Pharmacokinetics of Subcutaneous Injection of OCTA101 in Adult Patients With Severe Hemophilia A
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to SADRs
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SubQ8-01
Record Dates: First submitted 2019-07-18; First posted 2019-08-06 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Severe Hemophilia A
Keywords: Hemophilia A; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Factor VIII
MeSH Terms: conditions — Hemophilia A; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): 50 IU/kg (n=4): single-period investigation with a single sc dose of 50 IU/kg OCTA101 profiled up to 72 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 2, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  Interventions: Drug: OCTA101
- Cohort 2 (Experimental): 100 IU/kg (n=4): single-period investigation with a single sc dose of 100 IU/kg OCTA101 profiled up to 96 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 3, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  Interventions: Drug: OCTA101
- Cohort 3 (Experimental): 50 IU/kg (n=8): two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 4 and 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  Interventions: Drug: OCTA101
- Cohort 5 (Experimental): (n=4): Three-period investigation of single sc doses of 20, 40, and 60 IU/kg OCTA101 profiled up to 72 hours after dosing. Treatments were to be administered in fixed dose-ascending sequence.
  Interventions: Drug: OCTA101
- Cohort 6 (Experimental): (n=16): Following an initial 4 to 6-week run-in period with Nuwiq iv prophylaxis, >3-6 months daily prophylactic treatment with 12.5 IU/kg OCTA101 sc, then 25 IU/kg OCTA101 sc for a further 6-7 months (exact dosing depends on available vial sizes). In case of two spontaneous bleeding episodes, after having completed at least 3 months with 12.5 IU/kg OCTA101 daily treatment the individual treatment dose will be increased from 12.5 to 25 IU/kg. Site of administration (abdomen or thigh) to be chosen by the patient. A further treatment phase with 40 IU/kg OCTA101 will be discussed with the DMC, once results of earlier dosing phases are available.
  Interventions: Drug: OCTA101

INTERVENTIONS:
Drug: OCTA101 — OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).

SUMMARY:
This Phase 1/2 study will be a dose escalation study in adults in 5 cohorts (named cohorts 1, 2, 3, 5 and 6), with the main purpose to assess the safety of subcutaneous injection of OCTA101 (a human-cl rhFVIII and recombinant human von Willebrand Factor fragment dimer) in previously treated adult patients with severe hemophilia A. The study also aims to assess the pharmacokinetics (PK) characteristics, dose proportionality, and subcutaneous bioavailability of OCTA101 compared with intravenous administration of Nuwiq (Human-cl rh FVIII), in order to define the prophylactic treatment (dose and injection interval) that would result in protective trough levels of FVIII:C for future Phase 3 studies. Cohorts 1, 2, 3 and 5 will undergo a single injection of OCTA101, with cohorts 1, 2 and 3 proceeding to 3-month daily dosing prophylactic treatment for 3 months by Data Monitoring Committee recommendation. Cohorts 1 and 2 will undergo a further PK at the end of the daily injection period. A further cohort, cohort 6, will have an initial 4 to 6-week run-in treatment period with Nuwiq intravenous prophylaxis followed by 12.5 IU/kg OCTA101 subcutaneous daily prophylaxis for >3 up to 6-7 months.

ELIGIBILITY:
Inclusion Criteria:

1. Severe hemophilia A (<1% FVIII:C) as documented in medical records
2. Males ≥18 years of age
3. Subjects who have had ≥150 exposure days (EDs) with a FVIII product
4. Written informed consent for study participation obtained before undergoing any study specific procedures

Exclusion Criteria:

1. Previous participation in this trial
2. Use of an Investigational Medicinal Product within 30 days prior to the first OCTA101 injection
3. History of FVIII inhibitors titre ≥0.6 BU/mL defined by medical records
4. Inhibitors to FVIII (≥0.6 BU/mL) at screening measured by Nijmegen modified Bethesda method at central laboratory
5. Human immunodeficiency virus (HIV) positive subjects with a CD4+ count <200/mL
6. Clinically significant anemia at screening (hemoglobin <8 g/dL)
7. Presence of any significant comorbidity (at the discretion of the investigator) that might confound the interpretation of the study data and/or that might put the patient at undue risk by participating in the trial
8. Any coagulation disorder other than hemophilia A
9. AST or ALT levels >3 times the upper limit of normal
10. Creatinine >120 μmol/L
11. Platelet count <100,000 μL
12. BMI ≥30 kg/m²
13. For Cohort 6, patients with a positive LumiTope test at screening will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients only
Enrollment: 36 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Specialized Hospital for Active Treatment of Hematological Diseases EAD Clinic of Clinical Hematology, Sofia, Bulgaria

REFERENCES:
- [Background] Cannavo A, Valsecchi C, Garagiola I, Palla R, Mannucci PM, Rosendaal FR, Peyvandi F; SIPPET study group. Nonneutralizing antibodies against factor VIII and risk of inhibitor development in severe hemophilia A. Blood. 2017 Mar 9;129(10):1245-1250. doi: 10.1182/blood-2016-06-720086. Epub 2016 Dec 29. PMID 28034891
- [Background] Gibaldi M. (1991) Biopharmaceutics and Clinical Pharmacokinetics. 4th Edition, Lea and Febiger, Philadelphia, Appendix II.
- [Background] Liesner RJ, Abashidze M, Aleinikova O, Altisent C, Belletrutti MJ, Borel-Derlon A, Carcao M, Chambost H, Chan AKC, Dubey L, Ducore J, Fouzia NA, Gattens M, Gruel Y, Guillet B, Kavardakova N, El Khorassani M, Klukowska A, Lambert T, Lohade S, Sigaud M, Turea V, Wu JKM, Vdovin V, Pavlova A, Jansen M, Belyanskaya L, Walter O, Knaub S, Neufeld EJ. Immunogenicity, efficacy and safety of Nuwiq(R) (human-cl rhFVIII) in previously untreated patients with severe haemophilia A-Interim results from the NuProtect Study. Haemophilia. 2018 Mar;24(2):211-220. doi: 10.1111/hae.13320. Epub 2017 Aug 16. PMID 28815880
- [Background] Smith BP, Vandenhende FR, DeSante KA, Farid NA, Welch PA, Callaghan JT, Forgue ST. Confidence interval criteria for assessment of dose proportionality. Pharm Res. 2000 Oct;17(10):1278-83. doi: 10.1023/a:1026451721686. PMID 11145235
- [Background] Wagner JG (1975) Fundamentals of clinical pharmacokinetics. Drug Intelligence Publications, Inc. Hamilton, IL, USA

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 50 IU/kg (n=4): single-period investigation with a single sc dose of 50 IU/kg OCTA101 profiled up to 72 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 2, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 2: 100 IU/kg (n=4): single-period investigation with a single sc dose of 100 IU/kg OCTA101 profiled up to 96 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 3, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 3: 50 IU/kg (n=8): two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 6: Following an initial 4-6-week run-in period with Nuwiq iv prophylaxis, 6-month prophylactic treatment with 12.5 IU/kg OCTA101 sc daily was planned. Sixteen patients entered the Nuwiq iv run-in and 10 patients went on to receive OCTA101 12.5 IU/kg. The study was terminated before treatment could be completed.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Started | 4 | 4 | 8 | 4 | 16
Completed Initial PK Assessment | 4 | 4 | 8 | 4 | 0 (PK assessment not carried out in these patients)
Started Daily Prophylaxis With OCTA-101 | 4 | 4 | 8 | 0 (Prophylaxis not planned for this cohort) | 10
Completed 3-month Daily Prophylaxis With OCTA-101 | 4 | 2 | 0 | 0 | 10
Completed | 4 | 2 | 0 | 4 | 1
Not Completed | 0 | 2 | 8 | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- Cohort 6: (n≥16): following an initial 4-6-week run-in period with Nuwiq iv prophylaxis, 6-month prophylactic treatment with 12.5 IU/kg OCTA101 sc daily was planned. Sixteen patients entered the Nuwiq iv run-in and 10 patients went on to receive OCTA101 12.5 IU/kg. The study was terminated before treatment could be completed.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (7.35) | 40.5 (11.82) | 43.5 (12.78) | 29.5 (5.51) | 41.9 (12.37) | 38.8 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 4 | 8 | 4 | 16 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic or Latino | 4 | 4 | 8 | 4 | 16 | 36
Region of Enrollment [Number; unit: participants]
  Bulgaria | 4 | 4 | 8 | 4 | 16 | 36
BMI [Mean (Standard Deviation); unit: kg per m2] | 27.7 (2.79) | 27.1 (3.14) | 25.3 (3.89) | 27.8 (3.59) | 24.6 (5.03) | 26.6 (3.42)
Haemophilia joint health score [Mean (Standard Deviation); unit: units on a scale] — Haemophilia joint health score (HJHS) evaluates six index joints to produce a score between 0-124. The maximum score for an individual index joint is 20. Higher scores indicate worse joint health.
  units on a scale | 24.3 (19.65) | 27.8 (26.11) | 23.3 (12.61) | 16.3 (8.14) | 21.25 (11.38) | 23.0 (15.89)

OUTCOME MEASURES:

1. Primary Outcome: Patients Experiencing Adverse Events
Time Frame: Approximately 4 months; up to 11 months for cohort 6
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 2 | 1 | 0 | 3

2. Primary Outcome: Participants Experiencing Dose-limiting Toxicities (DLTs)
Description: Pre-defined DLTs for this study are: 1. Severe allergic reactions at least possibly related to study drug. 2. Severe vital organ toxicity at least possibly related to study drug that does not resolve to at least mild severity within 48 to 72 hours. 3. Any treatment-emergent severe toxicity at least possibly related to study drug other than the toxicities referenced in 2) that does not decrease to mild or resolve within 7 days
Time Frame: Approximately 4 months; up to 11 months for cohort 6
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Patients Experiencing Thromboembolic Events
Description: The definition of the cluster thromboembolic events was based on the standardised MedDRA query (SMQ) "Embolic and thrombotic events":
  Definition: Thrombotic disorders are diseases characterized by formation of a thrombus that obstructs vascular blood flow locally or detaches and embolizes to occlude blood flow downstream. Embolism is the sudden blocking of a vessel by a clot or foreign material which has been brought to its site of lodgment by the blood current. (Thrombo-)phlebitis is an inflammation of a vein (phlebitis) associated with thrombus formation (thrombosis).
  This SMQ includes 3 sub-SMQ:
  * Embolic and thrombotic events, venous (SMQ)
  * Embolic and thrombotic events, arterial (SMQ)
  * Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous (SMQ)
Time Frame: Approximately 4 months; up to 11 months for cohort 6
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Patients Experiencing Local Injection Site Reactions of Any Grade
Description: Investigator (and patient in case of home treatment) assessed local injection reactivity directly after injection and at 15 ± 5 min post-injection as per the ISO10999-10 standard:
  0=no skin reactivity;
  1. mild (subject is aware of the signs/symptoms, but finds it easily tolerated)
  2. moderate (discomfort enough to cause interference with usual activities)
  3. severe (subject is incapacitated and unable to work or participate in many or all usual activities).
Time Frame: Approximately 4 months; up to 11 months for cohort 6. Local injection site reactions were captured throughout the period where OCTA-101 was injected subcutaneously (sc).
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3: 50 IU/kg: two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 5: Three-period investigation of single sc doses of 20, 40, and 60 IU/kg OCTA101 profiled up to 72 hours after dosing. Treatments were to be administered in fixed dose-ascending sequence.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: Inhibitor Formation to FVIII
Description: Development of an inhibitor was defined as a neutralizing antibody value of greater than or equal to (>=) 0.6 Bethesda units per milliliter (BU/mL) identified and confirmed by a second test on an independent sample. In case of positive inhibitor results, inhibitor retesting using a second, separately drawn sample was to be performed, preferably within 15 days of becoming aware of the positive result. Both tests performed by the central laboratory using Nijmegen-modified Bethesda assay.
Time Frame: From first injection to 4 months after start of of daily injection (cohorts 1, 2 and 3), 4 weeks after last PK injection (cohort 5), monthly during the daily sc treatment period (cohort 6)
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 2 | 1 | 0 | 2

6. Secondary Outcome: Efficacy: Area Under the Concentration-time Curve (AUC) of FVIII:C
Description: Mean AUC of FVIII after PK injection of OCTA101 as measured by chromogenic assay.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: Cohort 5 data is given for 40 IU/kg dose. No PK data for cohort 6. For 1 patient in cohort 2, the measurable the levels of FVIII:C were very low and not evaluable by conventional non-compartmental PK
Measure: Mean (Standard Deviation); unit: IU*h/mL per IU/kg dosed
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
IU*h/mL per IU/kg dosed | 0.06265 (0.02606) | 0.05453 (0.01934) | 0.06558 (0.04452) | 0.0695 (0.0274) |

7. Secondary Outcome: Efficacy: Maximum Plasma Concentration (Cmax) of FVIII:C
Description: Maximum observed concentration of FVIII:C after PK injection of OCTA101 as measured by chromogenic assay.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: For 1 patient in cohort 2, the measurable the levels of FVIII:C were very low and not evaluable by conventional non-compartmental PK). Cohort 5 data is given for 40 IU/kg dose. No PK data for cohort 6.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
IU/mL | 0.082 (0.012) | 0.143 (0.065) | 0.074 (0.034) | 0.107 (0.014) |

8. Secondary Outcome: Efficacy: Time for Reaching Maximum Plasma Concentration (Tmax) of FVIII:C
Description: Time of occurrence of Cmax after PK injection of OCTA101 as measured by chromogenic assay.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
hours | 8.04 (0.06) | 18.92 (10.23) | 13.56 (6.49) | 11.11 (0.02) |

9. Secondary Outcome: In Vivo Recovery (IVR) of FVIII:C
Description: In vivo recovery (IVR) = dose-normalised and body weight-normalised maximum gain in FVIII:C (IU/dL per IU/kg)
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
IU/dL per IU/kg | 0.146 (0.021) | 0.132 (0.056) | 0.135 (0.058) | 0.233 (0.033) |

10. Secondary Outcome: Efficacy: Half-life (t1/2) of FVIII:C
Description: Apparent terminal log-linear half-life of FVIII:C after PK injection of OCTA101 as measured by chromogenic assay.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
hours | 22.74 (12.40) | 24.45 (6.92) | 26.59 (10.19) | 22.77 (4.88) |

11. Secondary Outcome: Efficacy: Mean Residence Time (MRT) of FVIII:C
Description: The average time at which the number of absorbed FVIII molecules reside in the body, after PK injection of OCTA101 as measured by chromogenic assay.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 0
hours | 37.91 (18.90) | 40.50 (3.86) | 43.08 (15.70) | 37.97 (7.99) |

12. Secondary Outcome: Efficacy: Area Under the Concentration-time Curve (AUC(0-tz)) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: Measurement of OCTA12 plasma concentrations using a validated ELISA in a central lab. Note: OCTA12 was not determined for cohort 6 regarding PK assessment.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Cohort 3: 50 IU/kg (n=8): two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 4 and 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5
Number analyzed (Participants) | 4 | 4 | 8 | 4
ng*h/mL | 3083.3 (701.3) | 7061.5 (3436.5) | 2897.9 (1049.2) | 1762.9 (589.9)

13. Secondary Outcome: Efficacy: Maximum Plasma Concentration (Cmax) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: as for outcome 12
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5
Number analyzed (Participants) | 4 | 4 | 8 | 4
ng/ml | 59.6 (11.69) | 95.8 (38.8) | 54.31 (19.25) | 32.95 (11.5)

14. Secondary Outcome: Efficacy: Time for Reaching Maximum Plasma Concentration (Tmax) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: as for outcome 12
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5
Number analyzed (Participants) | 4 | 4 | 8 | 4
hours | 71.46 (1.01) | 71.39 (19.22) | 68.15 (8.41) | 59.26 (13.71)

15. Secondary Outcome: Efficacy: In Vivo Recovery (IVR) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: In vivo recovery (IVR) = dose-normalised and body weight-normalised maximum gain in OCTA-12 (ug/dL per ug/kg).
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: The total of 20 participants were divided between their assigned cohorts.
Measure: Number; unit: ug/dL per ug/kg
Groups:
- In Vivo Recovery: Measure type: number Unit of Measure: ug/dL per ug/kg
Arm/Group | In Vivo Recovery
Number analyzed (Participants) | 20
ug/dL per ug/kg
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate IVR
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate IVR
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate IVR
  Cohort 5: number analyzed (Participants) | 4
  Cohort 5 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate IVR

16. Secondary Outcome: Efficacy: Half Life (t1/2) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: Measurement of OCTA12 plasma concentrations using a validated ELISA in a central lab. Note: t(1/2) could not be determined for OTCA12 as the OCTA12 concentrations had not yet declined during the observation time prior to prior to end of sampling period.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: The total of 20 participants were divided between their assigned cohorts.
Measure: Number; unit: hours
Groups:
- Half Life (t1/2): Measure type: number Unit of Measure: hours
Arm/Group | Half Life (t1/2)
Number analyzed (Participants) | 20
hours
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate t1/2
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate t1/2
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate t1/2
  Cohort 5: number analyzed (Participants) | 4
  Cohort 5 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate t1/2

17. Secondary Outcome: Efficacy: Mean Residence Time (MRT) of OCTA12 (a Recombinant Von Willebrand Factor Fragment Dimer)
Description: Note: MRT could not be determined for OCTA12 as the OCTA12 concentrations had not yet declined during the observation time prior to end of sampling period.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,3,5) or 96 hours (cohort 2)
Population: The total of 20 participants were divided between their assigned cohorts.
Measure: Number; unit: hours
Groups:
- Mean Residence Time (MRT): Measure type: number Unit of Measure: hours
Arm/Group | Mean Residence Time (MRT)
Number analyzed (Participants) | 20
hours
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate MRT
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate MRT
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate MRT
  Cohort 5: number analyzed (Participants) | 4
  Cohort 5 | NA — The time courses of the plasma concentrations of OCTA12 were not profiled for a sufficiently long time to observe a decline in the OCTA12 plasma concentrations and thus it was not possible to calculate MRT

18. Secondary Outcome: Efficacy: Total Annualized Bleeding Rate
Description: Total annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3 An estimated total annualized bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate for cohort 6.
Time Frame: The median (min, max) duration of daily sc treatment with OCTA101 in the 16 patients of cohort 1, 2 and 3 was 42 days (22, 93).
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: Annualized number of bleedings
Groups:
- Total Bleeding Rate: Measure type: number Unit of Measure: bleeding events per year
Arm/Group | Total Bleeding Rate
Number analyzed (Participants) | 26
Annualized number of bleedings
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

19. Secondary Outcome: Efficacy: Spontaneous Annualized Bleeding Rate
Description: Spontaneous annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3
  An estimated total spontaneous annualized bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate
Time Frame: as for outcome 18
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: Total bleeding events per year
Groups:
- Total Bleeding Rate: Measure type: number Unit of Measure: annualized number of bleedings
Arm/Group | Total Bleeding Rate
Number analyzed (Participants) | 26
Total bleeding events per year
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

20. Secondary Outcome: Efficacy: Total Annualized Treated Bleeding Rate
Description: Total annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3
  An estimated total annualized treated bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate.
Time Frame: as for outcome 18
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: bleeding events per year
Arm/Group | Total Bleeding Rate
Number analyzed (Participants) | 26
bleeding events per year
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

21. Secondary Outcome: Efficacy: Spontaneous Annualized Treated Bleeding Rate
Description: Spontaneous annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3.
  An estimated total spontaneous annualized treated bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate.
Time Frame: as for outcome 18
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: bleeding events per year
Groups:
- Total Bleeding Rates: Measure type: number Unit of Measure: annualized number of bleedings
Arm/Group | Total Bleeding Rates
Number analyzed (Participants) | 26
bleeding events per year
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

22. Secondary Outcome: Efficacy: Traumatic Annualized Bleeding Rate
Description: Traumatic annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3
  An estimated total traumatic annualized bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate.
Time Frame: as for outcome 18
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: Total bleeding events per year
Arm/Group | Total Bleeding Rate
Number analyzed (Participants) | 26
Total bleeding events per year
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

23. Secondary Outcome: Efficacy: Joint Annualized Bleeding Rate
Description: Joint annualized bleeding rate during daily subcutaneous treatment with OCTA101 for cohorts 1, 2 and 3.
  An estimated total joint annualized bleeding rate was calculated for cohorts 1,2 and 3. As these were estimated rates, there is only one value for each cohort with no measure of spread.
  As the study was terminated so soon, it was not considered accurate to extrapolate results to one year for annualized bleeding rate.
Time Frame: as for outcome 18
Population: The total of 26 participants were divided between their assigned cohorts.
Measure: Number; unit: Total bleeding events per year
Arm/Group | Total Bleeding Rate
Number analyzed (Participants) | 26
Total bleeding events per year
  Cohort 1: number analyzed (Participants) | 4
  Cohort 1 | 0
  Cohort 2: number analyzed (Participants) | 4
  Cohort 2 | 0
  Cohort 3: number analyzed (Participants) | 8
  Cohort 3 | 0
  Cohort 6: number analyzed (Participants) | 10
  Cohort 6 | NA — Due to study termination this outcome was not calculated for cohort 6.

24. Secondary Outcome: Efficacy: FVIII:C Trough and Peak Plasma Levels
Description: FVIII:C trough and peak plasma levels during daily dosing for cohorts 1, 2, 3 and 6
Time Frame: 3 months; maximally 6 months for cohort 6
Population: Not all patients in cohort 2 and 3 were analyzed at month 2 and 3 due to study termination. Only 3 patients were analyzed in cohort 6 at month 3 due to study termination. No PK analysis were performed for cohort 6.
Measure: Median (Full Range); unit: IU/mL
Groups:
- Cohort 1 Predose; Cohort 1 - 3 Hours; Cohort 1 - 6 Hours: 50 IU/kg (n=4): single-period investigation with a single sc dose of 50 IU/kg OCTA101 profiled up to 72 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 2, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 2 Predose; Cohort 2 - 3 Hours; Cohort 2 - 6 Hours: 100 IU/kg (n=4): single-period investigation with a single sc dose of 100 IU/kg OCTA101 profiled up to 96 hours after dosing in adult male patients with severe hemophilia A.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 3, alongside daily prophylactic dosing (40-60 IU/kg) for 3 months. In months 2 and 3 data could not be collected from all participants.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 3 Predose: 50 IU/kg (n=8): two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  The study was terminated before treatment could be completed, as a result, no data was collected in months 2 and 3.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
- Cohort 3 - 3 Hours; Cohort 3 - 6 Hours: 50 IU/kg (n=8): two-period investigation of a single iv dose of 50 IU/kg Human-cl rhFVIII (Nuwiq) profiled for up to 72 hours after dosing followed by sc dose of 50 IU/kg OCTA101 profiled up to 72 hours in adult male patients with severe hemophilia A.
  Treatments will be administered in fixed sequence, with Human-cl rhFVIII first.
  Following review of safety and tolerability data by Data Monitoring Committee, proceed with Cohort 5 alongside daily prophylactic dosing (40-60 IU/kg) for 3 months.
  The study was terminated before treatment could be completed, as a result, no data was collected in months 2 and 3.
- Cohort 6 Predose; Cohort 6 - 8 Hours: Following an initial 4-6-week run-in period with Nuwiq iv prophylaxis, 6-month prophylactic treatment with 12.5 IU/kg OCTA101 sc daily was planned. Sixteen patients entered the Nuwiq iv run-in and 10 patients went on to receive OCTA101 12.5 IU/kg. The study was terminated before treatment could be completed, so in month 3 data could not be collected from all participants.
Arm/Group | Cohort 1 Predose | Cohort 1 - 3 Hours | Cohort 1 - 6 Hours | Cohort 2 Predose | Cohort 2 - 3 Hours | Cohort 2 - 6 Hours | Cohort 3 Predose | Cohort 3 - 3 Hours | Cohort 3 - 6 Hours | Cohort 6 Predose | Cohort 6 - 8 Hours
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 8 | 16 | 16
IU/mL
  Start of daily treatment: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 8 | 10 | 10
  Start of daily treatment | 0.0035 [0.0035 to 0.0035] | 0.0210 [0.004 to 0.036] | 0.0375 [0.004 to 0.066] | 0.0058 [0.004 to 0.015] | 0.0160 [0.004 to 0.036] | 0.0245 [0.008 to 0.046] | 0.0090 [0.004 to 0.050] | 0.0405 [0.008 to 0.067] | 0.0645 [0.020 to 0.091] | 0.0035 [0.0035 to 0.0250] | 0.0170 [0.0035 to 0.0350]
  Month 0.5: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 8 | 9 | 10
  Month 0.5 | 0.1125 [0.099 to 0.172] | 0.1395 [0.112 to 0.193] | 0.1580 [0.126 to 0.207] | 0.0620 [0.013 to 0.196] | 0.1015 [0.015 to 0.261] | 0.1270 [0.010 to 0.290] | 0.1025 [0.044 to 0.547] | 0.1120 [0.065 to 0.490] | 0.1440 [0.070 to 0.514] | 0.0150 [0.0035 to 0.0310] | 0.0250 [0.0150 to 0.0450]
  Month 1: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 8 | 8 | 8 | 10 | 10
  Month 1 | 0.1885 [0.180 to 0.288] | 0.1995 [0.195 to 0.310] | 0.2175 [0.216 to 0.293] | 0.0465 [0.004 to 0.088] | 0.0515 [0.004 to 0.104] | 0.0615 [0.009 to 0.133] | 0.1080 [0.035 to 0.272] | 0.1250 [0.056 to 0.275] | 0.1610 [0.072 to 0.261] | 0.0185 [0.0035 to 0.0360] | 0.0280 [0.0035 to 0.0690]
  Month 2: number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 0 | 0 | 0 | 10 | 10
  Month 2 | 0.1510 [0.090 to 0.169] | 0.1920 [0.161 to 0.236] | 0.2155 [0.190 to 0.296] | 0.0120 [0.004 to 0.089] | 0.0110 [0.004 to 0.103] | 0.0100 [0.004 to 0.106] |  |  |  | 0.0190 [0.0035 to 0.0380] | 0.0325 [0.0035 to 0.0510]
  Month 3: number analyzed (Participants) | 4 | 4 | 4 | 2 | 2 | 2 | 0 | 0 | 0 | 3 | 3
  Month 3 | 0.1645 [0.102 to 0.208] | 0.1995 [0.149 to 0.290] | 0.2250 [0.193 to 0.227] | 0.0655 [0.014 to 0.117] | 0.0698 [0.004 to 0.136] | 0.0775 [0.008 to 0.147] |  |  |  | 0.0120 [0.0035 to 0.0290] | 0.0230 [0.0160 to 0.0330]

25. Secondary Outcome: Efficacy: Efficacy of Treatment of Bleeding Episodes Using Score (4-point).
Description: Score (4-point) to assess the efficacy of treatment of bleeding episodes with Human-cl rhFVIII. Treatment efficacy will be assessed using predefined criteria to score either 'Excellent', 'Good', 'Moderate' or 'None'. All efficacy ratings assessed as either 'excellent' or 'good' will be considered 'successfully treated'.
Time Frame: 5 days to approximately 11 months
Reporting Status: Not Posted

26. Secondary Outcome: Safety: Antibody Formation to OCTA12
Description: Samples were checked for the presence of antibodies to OCTA12 by using a validated ELISA in a central lab.
Time Frame: From 0 hours (pre-dose) to 72 hours (cohorts 1,2,3,5) or 96 hours (cohort 2).
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Safety: OCTA12 Plasma Levels
Description: OCTA12 plasma levels during daily dosing (cohorts 1, 2, 3 and 6).
Time Frame: 3 months; maximally 6 months for cohort 6
Reporting Status: Not Posted

28. Secondary Outcome: Safety: Change in Hemoglobin
Description: Number of Participants with changes in hemoglobin levels that were considered as Adverse Events.
Time Frame: 5 days to approximately 11 months. All routine lab parameters and vital signs were measured at various times, until end of PK and also monthly during daily prophylaxis.)
Reporting Status: Not Posted

29. Secondary Outcome: Safety: Change in Alanine Aminotransferase (ALT)
Description: Alanine aminotransferase (ALT) compared to baseline, measured in U/L. Number of Participants with changes in ALT that were considered as Adverse Events.
Time Frame: as for outcome 28
Reporting Status: Not Posted

30. Secondary Outcome: Safety: Change in Aspartate Transaminase (AST)
Description: Aspartate transaminase (AST) compared to baseline, measured in U/l. Number of Participants with changes in AST that were considered as Adverse Events.
Time Frame: 5 days to approximately 11 months
Reporting Status: Not Posted

31. Secondary Outcome: Patients With Changes to Vital Signs
Description: Vitals signs changes from baseline, reported as AEs. Number of Participants with changes to vital signs that were considered as Adverse Events.
Time Frame: 5 days to approximately 11 months
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Patients With Changes in Physical Examination Results
Description: Number of Participants with changes to their physical examination results from baseline that were considered as Adverse Events
Time Frame: 5 days to approximately 11 months
Population: The population included all patients who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 4 | 4 | 8 | 4 | 10
Participants | 0 | 2 | 1 | 0 | 3

ADVERSE EVENTS:
Time Frame: Approximately 4 months; up to 11 months for cohort 6
Description: An adverse event is any untoward medical occurrence in a study patient receiving an IMP and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not related to the IMP.
Groups:
- Cohort 6: (n≥16): following an initial 4-6-week run-in period with Nuwiq iv prophylaxis, 6-month prophylactic treatment with 12.5 IU/kg OCTA101 sc daily was planned. Sixteen patients entered the Nuwiq iv run-in and 10 patients went on to receive OCTA101 12.5 IU/kg. The study was terminated before treatment could be completed in all but 1 patient.
  OCTA101: OCTA101 is composed of OCTA8 (human-cl rhFVIII - Nuwiq Intermediate 2 Q-Eluate) and OCTA12 (recombinant human VWF fragment dimer).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 0/8 | 0/4 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 1/8 | 0/4 | 2/16
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 0/8 | 0/4 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=8) | Cohort 5 (N=4) | Cohort 6 (N=16)
Anti Factor VIII antibody positive (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spontaneous hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Retroperitoneal hematoma
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=8) | Cohort 5 (N=4) | Cohort 6 (N=16)
Injection site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Roseolovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT04046848/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT04046848/SAP_001.pdf